CLINICAL TRIAL: NCT03404284
Title: Assessment of Family Planning and Immunization Service Integration in Malawi
Status: Completed | Type: Observational
Sponsor: Jhpiego (Other)
Collaborators: John Snow, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: IRB00007595
Record Dates: First submitted 2018-01-11; First posted 2018-01-19 (Actual); Last update posted 2018-01-19 (Actual); Status verified 2018-01

CONDITIONS: Contraception; Contraceptive Usage; Contraception Behavior; Infant, Newborn, Diseases
Keywords: Immunization
MeSH Terms: conditions — Contraception Behavior; Infant, Newborn, Diseases | interventions — Family Planning Services

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Intervention facilities: Includes 43 health facilities and their associated outreach sites
  Interventions: Behavioral: Family planning and infant immunization service integration

INTERVENTIONS:
Behavioral: Family planning and infant immunization service integration — The approach involved integration of services through health surveillance assistant (HSA) outreach as well as through the health facility platform. The HSAs provided door to door FP services in their designated communities as well as provided integrated FP and Immunisation services at village clinics and outreach sessions. At outreach sessions, mothers were offered both routine infant immunization and family planning services (pills, condoms, injectables plus referrals for other methods). At health facilities, mothers who sought routine infant immunization services were offered same-day family planning services and those who seek family planning services are also screened for infant immunization schedule completion / need for infant immunization services. HSAs and health facility providers were trained on FP-immunization service integration and were monitored through regular supportive supervision visits.

SUMMARY:
This is a mixed methods process evaluation of a programmatic intervention to integrate family planning and immunization services at health facilities and through outreach services in Dowa and Ntchisi districts of Malawi. The study involved qualitative methods (in depth interviews and focus group discussions with service providers, mothers and fathers of infants <1 year, and supervisors and program managers) as well as secondary analysis of service statistics for family planning and immunization services and of supervision reports.

ELIGIBILITY:
Inclusion Criteria:

* All health facilities and associated outreach sites in Ntchisi and Dowa districts implementing the integrated approach with support from the USAID-funded Maternal and Child Survival Program

Exclusion Criteria:

* All health facilities and associated outreach sites not implementing the integrated approach with support from the USAID-funded Maternal and Child Survival Program

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: 43 health facilities and associated outreach sites in Ntchisi and Dowa districts of Malawi
Sampling Method: Non-Probability Sample
Enrollment: 43 (Actual)
Dates: Start 2016-06 (Actual); Primary Completion 2017-09 (Actual); Study Completion 2017-09 (Actual)

PRIMARY OUTCOMES:
Number of modern family planning users | June 2016 through September 2017 (we also collected pre-intervention data from January to May 2016)
Number of Penta 1 doses administered | June 2016 through September 2017 (we also collected pre-intervention data from January to May 2016)
Number of Penta 3 doses administered | June 2016 through September 2017 (we also collected pre-intervention data from January to May 2016)

IPD SHARING:
Plan to Share IPD: No